CLINICAL TRIAL: NCT05989087
Title: The Underestimated Utility of Resting-state Gamma Oscillations: Both Increase and Decrease of Gamma Discriminates Early-onset Alzheimer's Disease Patients From Healthy Individuals
Brief Title: The Resting-state EEG Gamma Oscillations in Alzheimer's Disease
Acronym: EEG
Status: Completed | Type: Observational
Sponsor: Görsev Yener, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Görsev Yener, MD, PhD, Clinical Professor, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: DokuzEU EEG
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Alzheimer's disease; Gamma activity; Resting-state EEG; Discriminative power; MRI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early-onset Alzheimer's disease: Patients were recruited from the outpatient memory clinics of the Department of Neurology, Dokuz Eylül University Hospital. The patient group was diagnosed by an expert neurologist, according to the National Institute on Aging-Alzheimer's Association diagnostic criteria for Alzheimer's disease
  Interventions: Diagnostic Test: CSF
- Healthy controls: Age-and gender-matched healthy volunteers were recruited via advertisements and word-of-mouth.

INTERVENTIONS:
Diagnostic Test: CSF — Early-onset Alzheimer's disease patients underwent routine laboratory tests to obtain CSF samples. Also, all participants underwent structural MRI examinations and neuropsychological tests.
  Other Names: MRI; Neuropsychological tests
  Groups: Early-onset Alzheimer's disease

SUMMARY:
The literature suggests a strong association between amyloid accumulation and gamma alterations, emerging gamma activity as a biomarker candidate for Alzheimer's pathology. The present study aims to investigate resting-state gamma activity changes in Cerebrospinal fluid (CSF)-proven early-onset Alzheimer's disease (EOAD) patients with a holistic approach that employs structural and functional brain neuroimaging techniques, and neuropsychological aspects.

DETAILED DESCRIPTION:
This cross-sectional study included 24 drug-naive CSF-proven EOAD patients and age-, sex, and education-matched healthy controls. All participants underwent a detailed neuropsychological evaluation, resting-state electroencephalography (EEG) recording, and Magnetic Resonance Imaging (MRI). Gamma power and coherence were measured in total gamma (30-48 Hz), gamma-1 (30-35 Hz), gamma-2 (35-40 Hz), and gamma-3 (40-48 Hz) frequency bands. Gray matter volumes were extracted for 54 regions of interest (ROIs) and compared between groups. Discriminant analysis was performed to determine the classification accuracy of gamma activity for EOAD. Finally, correlations between CSF, neuropsychological tests, EEG, and MRI measures were explored.

ELIGIBILITY:
Inclusion Criteria:

* For all participants: Age < 65
* For EOAD patients: Meeting National Institute on Aging-Alzheimer's Association diagnostic criteria.
* For healthy controls: Mini-Mental State Examination (MMSE) >25 Instrumental Activities of Daily Living Scale (IADL) = 8

Exclusion Criteria:

* For EOAD patients: MMSE > 24 Geriatric depression scale (GDS) > 14 Having treatment with antipsychotics and comorbidities that may affect cognitive abilities.
* For healthy controls: Having neurological and/or cognitive abnormalities Having a history of neurological, psychiatric, or systemic disorders, and alcohol/drug abuse. GDS > 14
* For all participants: Having neurological (other than AD) or any other serious disease (cancer, systemic disease)

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The present study included a retrospective investigation of EEG and MRI data. The total sample for the study consisted of 24 early-onset Alzheimer's disease patients and 24 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2016-01-02 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
EEG | Day 2
  The resting state EEG recordings were acquired using Easy-Cap comprising 30 Ag/AgCl electrodes placed according to the international 10-20 system. Coherence and maximum peak power of the total gamma (30-48 Hz) and sub-gamma bands [gamma-1 (30-35 Hz), gamma-2 (35-40 Hz), and gamma-3 (40-48 Hz)] were measured for each participant.

SECONDARY OUTCOMES:
Correlation Analysis | 3 months
  Correlations between CSF, neuropsychological tests (NPT), EEG, and MRI measures were investigated.
Discriminant Analysis | 3 months
  The discriminative power of gamma measures (power and coherence) was investigated with discriminant analysis (DA).
MRI | Day 1
  Participants underwent structural magnetic resonance imaging on a Philips Achieva 1.5 Tesla scanner. The gray matter volumes were obtained from the 3D-T1 weighted Turbo field echo (TFE) sequence (TR: 9ms, Time to Echo (TE): 4ms, Field-of-view (FOV): 240mm, matrix: 256, slice thickness: 1mm, numbers of signal averages (NSA): 1). The images were segmented into gray matter, white matter, and CSF with the default parameters of the CAT12 segmentation function. Only the gray matter calculations were compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir University of Economics, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the contact person, upon reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT05989087/Prot_SAP_000.pdf